CLINICAL TRIAL: NCT03251430
Title: Assessment of Bone Microstructure by Using High-resolution Peripheral Quantitative Computed Tomography in Long Courses After Gastrectomy : a Prospective Observational Study
Brief Title: Bone Microstructure by Using HR-pQCT in Long Courses After Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kobayashi Shinichiro (Other)
Responsible Party: Sponsor-Investigator, Kobayashi Shinichiro, Principal Investigator in department of Surgery, Nagasaki University
Organization: Nagasaki University (Other)
Other Study IDs: 17061943
Record Dates: First submitted 2017-08-07; First posted 2017-08-16 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Osteoporosis; Sarcopenia; Gastric Cancer
MeSH Terms: conditions — Osteoporosis; Sarcopenia; Stomach Neoplasms | interventions — Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Protein
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control group: 38 patients without gastrectomy , who are similar background in other group, are collected from date Pathologic analysis of primary osteoporosis: investigating age and osteoporosis related changes of bone microstructure by using HR-pQCT (UMIN000023535)
- Distal Gastrectomy (DG) group: 38 patients with distal gastrectomy due to gastric cancer before no more than 5 years
  Interventions: Procedure: gastrectomy
- Total Gastrectomy (TG) group: 38 patients with distal gastrectomy due to gastric cancer before no more than 5 years
  Interventions: Procedure: gastrectomy

INTERVENTIONS:
Procedure: gastrectomy — Distal gastrectomy, Total gastrectomy
  Groups: Distal Gastrectomy (DG) group; Total Gastrectomy (TG) group

SUMMARY:
Osteoporosis after gastrectomy, which is characterized by both the loss of bone mass and the deterioration of bone architecture, is a serious complication in the long course after gastrectomy. The aim of the present study was to evaluate osteoporosis by using high-resolution peripheral quantitative computed tomography (HR-pQCT) in the long course after gastrectomy. In total gastrectomy and distal gastrectomy groups, at least 5 years should have elapsed since gastrectomy.

DETAILED DESCRIPTION:
The patients after gastrectomy loss appetite and decrease the weight. Total gastrectomy especially cause severe sarcopenia and metabolic change. Osteoporosis after gastrectomy, which is characterized by both the loss of bone mass and the deterioration of bone architecture, is a serious complication in the long course after gastrectomy. The primary tools for assessing volumetric density and bone structure are quantitative computed tomography (QCT) and more recently, high-resolution peripheral quantitative computed tomography (HR-pQCT). However the validation of osteoporosis with HR-pQCT in the long course after gastrectomy remain elusive. The aim of the present study was to evaluate osteoporosis by using HR-pQCT in the long course after gastrectomy. In total gastrectomy and distal gastrectomy groups, at least 5 years should have elapsed since gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* At least 5 years have elapsed since DG or TG due to gastric cancer
* Provide signed informed consent

Exclusion Criteria:

* pregnancy
* Current use of the following osteoporosis agents; Teriparatide, Denosumab, and bisphosphonate
* Hyperthyroidism
* Hyperparathyroidism
* Present malignancy (except in situ carcinoma)
* Any condition that required chronic (greater than three months cumulative and greater than 5 mg/day) glucocorticoid therapy
* Other diseases which affect bone metabolism
* Any disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or comply with study procedures
* Received > 3 months (or equivalent) of osteoporosis treatment
* Currently enrolled in or has not yet completed at least 1 month since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s).

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Japanese
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparing bone microstructure in control, DG, and TG groups | day1
  volumetric bone mineral density

SECONDARY OUTCOMES:
Comparing bone microstructure with sarcopenia | day1
  Correlation between bone mineral density in HR-pQCT and cross-sectional area of the abdominal psoas major muscle
Comparing bone microstructure with serum biomarkers of osteoporosis | day1
  Correlation between bone mineral density in HR-pQCT and biomarkers (25-hydroxyvitaminD, calcium, iPTH, P1NP, ICTP, TRACP5b)
Comparing bone microstructure with dual-energy X-ray absorptiometry | day1
  Correlation of bone mineral density between HR-pQCT and DXA
Comparing bone microstructure with quality of life (QOL-C30) | day1
  Patients will be asked to complete a short debriefing questionnaire covering questions (QOL-C30)
Comparing bone microstructure with quality of life (BDHQ) | day1
  Patients will be asked to complete a short debriefing questionnaire covering questions ( BDHQ)
Comparing bone microstructure with quality of life (FRAX) | day1
  Patients will be asked to complete a short debriefing questionnaire covering questions (FRAX)

CONTACTS AND LOCATIONS:
Overall Officials: Shinichiro Kobayashi, MD, Principal Investigator — Department of Surgery, Nagasaki University Graduate School of Biomedical Sciences,
Locations (1):
- Nagasaki University Hospital, Nagasaki, Japan

IPD SHARING:
Plan to Share IPD: No